CLINICAL TRIAL: NCT01268150
Title: A Phase 2, Multicenter, Single-Arm Study of Single-Agent Eribulin Mesylate as First-Line Therapy for Locally Recurrent or Metastatic Human Epidermal Growth Factor Receptor Two (HER2) Negative Breast Cancer
Brief Title: A Study of Single-Agent Eribulin Mesylate as First-Line Therapy for Locally Recurrent or Metastatic Human Epidermal Growth Factor Receptor Two (HER2) Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-206
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2016-06

CONDITIONS: Locally Recurrent; Metastatic Breast Cancer ( HER2 Negative)
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Eribulin mesylate

INTERVENTIONS:
Drug: Eribulin mesylate — Eribulin mesylate 1.4 mg/m2 will be administered as an intravenous (IV) infusion (over 2 to 5 minutes) on Days 1 and 8 of each 3-week cycle.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of single-agent eribulin mesylate for first-line treatment of subjects with locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, Phase 2 trial to assess the efficacy and safety of single-agent eribulin mesylate for first-line treatment of subjects with locally recurrent or metastatic human epidermal growth factor receptor (HER2)-negative breast cancer. A total of 52 adult female subjects will be enrolled and treated with eribulin mesylate (1.4 mg/m2 as an intravenous [i.v.] infusion over 2 to 5 minutes on Days 1 and 8 of each 3-week cycle).

ELIGIBILITY:
Key Inclusion Criteria

Females age 18 years or older at the time of informed consent

Have histologically or cytologically proven adenocarcinoma of the breast

Subjects with locally recurrent or metastatic disease with at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors

(RECIST) criteria v 1.1

Human epidermal growth factor receptor (HER2)-negative disease as determined by fluorescence in situ hybridization (FISH) or 0 or 1+ by immunohistochemical (IHC) staining.

Life expectancy of greater than 24 weeks

Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) of 0, 1 or 2

At least 12 months since prior neoadjuvant or adjuvant chemotherapy

At least 2 weeks since prior radiotherapy or endocrine therapy, with complete recovery from the effects of these interventions

Adequate renal function

Adequate bone marrow function

Adequate liver function

Key Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from participation in this study:

Prior chemotherapy, biologic therapy, or investigational therapy for locally recurrent or metastatic breast cancer

Subjects who have had a prior malignancy other than carcinoma in situ of the cervix or nonmelanoma skin cancer

Prior exposure of greater than 360 mg/m2 doxorubicin or liposomal doxorubicin, greater than 120 mg/m2 mitoxantrone, greater than 90 mg/m2 idarubicin, or greater than720 mg/m2 epirubicin

Inflammatory breast cancer

Clinically significant cardiovascular impairment

Subjects with known CNS disease are not eligible, except for those with treated brain metastasis.

Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring the use of oxygen

Currently pregnant or breast-feeding.

Subjects with pre-existing Grade 3 or 4 neuropathy. Any peripheral neuropathy must recover to Grade 2 before enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Misir, Study Director — Eisai Inc.
Locations (17):
- United States (17):
  - University of Miami, Miami, Florida
  - Augusta Oncology Associates, Augusta, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Missouri Cancer Associates, Columbia, Missouri
  - Hematology Oncology Centers of Northern Rockies, Billings, Montana
  - New York Oncology Hematology, P.C., Albany, New York
  - Weill Cornell Medical Center, New York, New York
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - The West Clinic, Memphis, Tennessee
  - Texas Oncology- Bedford, Bedford, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology- Tyler, Tyler, Texas
  - Columbia Basin Hematology and Oncology, Kennewick, Washington

REFERENCES:
- [Derived] McIntyre K, O'Shaughnessy J, Schwartzberg L, Gluck S, Berrak E, Song JX, Cox D, Vahdat LT. Phase 2 study of eribulin mesylate as first-line therapy for locally recurrent or metastatic human epidermal growth factor receptor 2-negative breast cancer. Breast Cancer Res Treat. 2014 Jul;146(2):321-8. doi: 10.1007/s10549-014-2923-9. Epub 2014 Apr 4. PMID 24699910

RESULTS

PARTICIPANT FLOW:
Groups:
- Eribulin Mesylate: Eribulin mesylate at 1.4 mg/m^2 was administered as an intravenous (IV) infusion over 2 to 5 minutes on Days 1 and 8 of each 3-week cycle.
Period: Treatment Phase
Arm/Group | Eribulin Mesylate
Started | 56
Completed | 28
Not Completed | 28
Not completed — Progression of disease | 18
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3
Not completed — Other | 4
Period: Extension Phase
Arm/Group | Eribulin Mesylate
Started | 28 (28 participants discontinued study drug in Treatment Phase so did not enter the Extension Phase)
Treatment Ongoing at Data Cutoff Date | 1
Completed | 1
Not Completed | 27
Not completed — Adverse Event | 3
Not completed — Disease progression | 18
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least one dose of study drug.
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of participants with best overall response (BOR) of confirmed complete response (CR) or partial response (PR), based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Targeted lesions were assessed by computed tomography (CT) and magnetic resonance imaging (MRI) which were then assessed by the investigator based on RECIST. CR was defined as the disappearance of all target lesions. PR was defined as at least 30% decrease in the sum of diameters of target lesions, taking as reference baseline sum diameters. Possible CR and PR had to be confirmed no fewer than 4 weeks after the initial response assessment. A brain and bone scan was performed by CT/MRI within 1 week after confirmation of a response to ensure no new metastases. To be assigned a status of CR or PR, changes in tumor measurements had to be confirmed by repeat evaluations, to be performed not fewer than 4 weeks after the response criteria were first met. ORR = CR + PR
Time Frame: Cycle 1 (Day 1) until first evidence of disease progression, assessed up to the data cutoff date (30 Aug 2013) up to 2.5 years
Population: Full analysis set included all participants who received at least one dose of eribulin mesylate.
Measure: Number; unit: Percentage of participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 56
Percentage of participants | 28.6

2. Secondary Outcome: Time to First Response (CR or PR)
Description: Time to first response was defined for participants whose BOR was a CR or PR. Analysis was based on the Kaplan-Meier estimated number of months to CR or PR. This statistical analysis method measures the effect of study drug on CR or PR.
Time Frame: Treatment Phase (Day 1 Cycle 1) to earliest date of confirmed objective response (CR or PR), assessed up to the data cutoff date (30 Aug 2013) up to 2.5 years
Population: Full analysis set included all participants who received at least one dose of eribulin mesylate and were determined to be responders (CR or PR) to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 16
Months | 1.4 [1.22 to 2.66]

3. Secondary Outcome: Duration of Response
Description: Duration of response was measured for participants who were responders only, had attained a BOR that was CR or PR. The duration of response was measured from time that response criteria for CR or PR (whichever was recorded first) were first met until the date that progressive disease (PD) or death from any cause was first objectively documented. Participants who did not have PD were censored on the day of their last tumor assessment. Duration of response was summarized for the responders using Kaplan-Meier estimation method. This statistical analysis method measures the effect of study drug on the length of response time.
Time Frame: First date of CR or PR to PD or Death from any cause, assessed up to the data cutoff date (30 Aug 2013) up to 2.5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 16
Months | 5.8 [4.67 to 10.55]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of the first dose of study drug until the date of first documentation of PD or date of death from any cause, whichever occurred first. Participants who died without reported PD were considered to have progressed on the day of their death. Participants who were lost to follow-up or alive and without reported PD at the end of study were censored on the date of their last tumor assessment. Participants without evidence of PD upon discontinuation of study drug during the Extension Phase returned to the clinic for disease evaluation and PFS calculation every 12 weeks until PD was documented. PFS was analyzed using Kaplan-Meier product-limit estimates. This statistical analysis method measures the effect of study drug on PFS.
Time Frame: Treatment Phase (Day 1 Cycle 1) to date of progressive disease or death, whichever occurred first, assessed up to the data cutoff date (30 Aug 2013) up to 2.5 years
Population: Full analysis set included all participants who received at least one dose of eribulin mesylate.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 56
Months | 6.8 [4.44 to 7.59]

5. Other Pre Specified Outcome: To Assess the Incidence of Adverse Events (AEs) of Eribulin Mesylate
Description: Treatment-emergent adverse events (TEAEs) were defined as AEs that emerged during treatment, having been absent at pretreatment, and occurring within 30 days of the last dose of study treatment, or if they were present prior to the first dose administration and increased in severity during the study. For each AE a participant with two or more TEAEs in that category were counted only once. TEAEs were considered related if the relationship of the event to study drug was possibly or probably related. Serious adverse events (SAEs) were defined as any untoward medical experience that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, persistent or significant disability/incapacity, or was a congenital anomaly/birth defect. Safety information will be summarized with adverse events. AEs were graded on a five-point scale according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Baseline until End of Treatment (within 21 days of last dose), assessed up to the data cutoff date (30 Aug 2013) up to 2.5 years
Population: Safety Analysis Set population included all participants who received at least one dose of study drug and had at least one postbaseline safety assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 56
Percentage of participants
  TEAEs | 100.0
  Treatment-related TEAEs | 100.0
  Serious TEAEs | 30.4
  Treatment-related Serious TEAEs | 8.9
  TEAEs leading to withdrawl of study drug | 10.7
  TEAEs leading to dose reduction | 35.7

ADVERSE EVENTS:
Time Frame: All Treatment-Emergent Adverse events (TEAEs) were collected and followed from the time the participant signed the informed consent form (ICF) until 30 days after discontinuation of study drug or resolution. Participants were followed for up to 2.5 years.
Description: Safety Analysis Set population included all participants who received at least one dose of study drug and had at least one postbaseline safety assessment. AEs were graded on a five-point scale according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. AEs rated as Grade 4 or 5 were considered serious.
Arm/Group | Eribulin Mesylate
Serious Adverse Events (participants affected / at risk) | 17/56
Other Adverse Events (participants affected / at risk) | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=56)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Pericardial effusion (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Spinal cord paralysis (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=56)
Anaemia (Blood and lymphatic system disorders) | 21
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 19
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 40
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Angina Pectoris (Cardiac disorders) | 2
Electrocardiogram QT prolonged (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1
Middle ear effusion (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Abnormal sensation in eye (Eye disorders) | 1
Cataract (Eye disorders) | 3
Dry Eye (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 7
Visual Impairment (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 5
Abdominal Pain Lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 4
Anal haemorrhage (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 20
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 19
Diverticulum intestinal (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 5
Food poisoning (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 33
Oral disorder (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Rectal fissure (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Salivary gland enlargement (Gastrointestinal disorders) | 1
Salivary gland mass (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 6
Tongue discolouration (Gastrointestinal disorders) | 1
Tooth deposit (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 14
Asthenia (General disorders) | 3
Axillary pain (General disorders) | 1
Catheter site erythema (General disorders) | 1
Catheter site inflammation (General disorders) | 2
Catheter site pain (General disorders) | 1
Catheter site rash (General disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 36
Gait disturbance (General disorders) | 2
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 2
Mucosal inflammation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema Peripheral (General disorders) | 11
Pain (General disorders) | 2
Pyrexia (General disorders) | 10
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Candidiadis (Infections and infestations) | 2
Catheter Site infection (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Pleural infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 11
Vaginal infection (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood glucose increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Helicobacter test positive (Investigations) | 1
International normalised ratio increased (Investigations) | 2
Liver function test abnormal (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Platelet count increased (Investigations) | 1
Prothrombin time prolonged (Investigations) | 1
Weight decreased (Investigations) | 9
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
White blood cell count increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Fluid retention (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Bunion (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2
Pubic pain (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ageusia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Balance Disorder (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 9
Head discomfort (Nervous system disorders) | 1
Headache (Nervous system disorders) | 13
Hypoaesthesia (Nervous system disorders) | 3
Hypogeusia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 2
Peroneal nerve palsy (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Spinal cord paralysis (Nervous system disorders) | 1
Peripheral Neuropathy (Nervous system disorders) | 34
Neuropathy peripheral (Nervous system disorders) | 26
Paraesthesia (Nervous system disorders) | 4
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 12
Affect lability (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 6
Disorientation (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 8
Mental status changes (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 9
Hydronephrosis (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 3
Pelvic pain (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 47
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 3
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 5
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 5
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Lymphoedema (Vascular disorders) | 2
Pallor (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 2
Thrombophlebitis superficial (Vascular disorders) | 1
Dysarthria (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No